CLINICAL TRIAL: NCT05569577
Title: An Open-labeled Prospective Randomized Controlled Trial on the Effect of Different Regimens for Luteal Phase Support on Pregnancy Outcomes in Patients With Idiopathic Hypogonadotropic Hypogonadism
Brief Title: An Open Labeled RCT on the Effect of Additional hCG Injection for LPS on Pregnancy Outcomes in IHH Patients
Acronym: LPS-IHH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhang Wei, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FudanU2022-08-18
Record Dates: First submitted 2022-10-02; First posted 2022-10-06 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Luteal Phase Deficiency; Luteal Phase Support; Idiopathic Hypogonadotropic Hypogonadism
Keywords: Luteal phase deficiency; Idiopathic hypogonadotropic hypogonadism
MeSH Terms: conditions — Idiopathic Hypogonadotropic Hypogonadism | interventions — Estrogens; Dydrogesterone

STUDY DESIGN:
Intervention Model Description: We have two cohorts in the current study and patients are randomly assigned to either cohort of additional hCG injection or not.
Masking Description: In the current study, none of patients, investigators and designers is marked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional hCG injection (Experimental): An additional hCG injection of 2000-5000IU would be performed 48 hours following routine hCG trigger on the basis of supplementation of estrogen and dydrogesterone in IHH patients.
  Interventions: Drug: Additional hCG injection; Drug: estrogen and dydrogesterone
- No additional hCG injection (Placebo Comparator): Only estrogen and dydrogesterone would be given for luteal phase support in IHH patients.
  Interventions: Drug: estrogen and dydrogesterone

INTERVENTIONS:
Drug: Additional hCG injection — An additional hCG injection of 2000-5000IU would be given 48 hours following routine hCG trigger and ovulation for LPS on the basis of supplementation of estrogen and dydrogesterone.
  Arms: Additional hCG injection
Drug: estrogen and dydrogesterone — estrogen and dydrogesterone

SUMMARY:
Luteal phase deficiency (LPD) accounts for most failures of assistant artificial reproduction (ART) and early pregnancy loss for patients with idiopathic hypogonadotropic hypogonadism (IHH). Luteal phase support (LPS) is one of the indispensable interventions in ART treatments for IHH patients, which includes progestin, estrogen, human chorionic gonadotropin (hCG), and GnRH agonists (GnRHa). We aim to verify additional hCG injection 48 hours following routine hCG trigger and ovulation for LPS on the basis of supplementation of estrogen and dydrogesterone could improve clinical pregnancy rate, cumulative pregnancy rate, live birth rate and the prevalence of early pregnancy loss and ovarian hyperstimulation syndrome (OHSS) by an open labeled, prospective, and randomized clinical trial (RCT) in IHH patients in a single center.

DETAILED DESCRIPTION:
Idiopathic hypogonadotropic hypogonadism (IHH) is a congenital disease caused by a variety of gene variants leading to dysfunction in the secretion of hypothalamic gonadotropin-releasing hormones (GnRHs), with a prevalence of 1:125 000 in females. Girls with IHH often suffer from lack of puberty onset, amenorrhea and infertility, complicated with psychological problems such as depression and anxiety, due to delayed diagnosis and inappropriate treatment. Luteal phase deficiency (LPD) accounts for most failures of assistant artificial reproduction (ART) and early pregnancy loss for IHH patients. We have reported a severe LPD during the early trimester in a case with secondary HH following craniopharyngioma resection and speculated similar LPD happen in IHH patients complicated with low clinical pregnancy rate and live birth rate. Therefore, luteal phase support (LPS) is one of the indispensable interventions in ART treatments for IHH patients, which includes progestin, estrogen, human chorionic gonadotropin (hCG), and GnRH agonists (GnRHa). We aim to verify additional hCG injection 48 hours following routine hCG trigger and ovulation for LPS on the basis of supplementation of estrogen and dydrogesterone could improve clinical pregnancy rate, cumulative pregnancy rate, live birth rate and the prevalence of early pregnancy loss and ovarian hyperstimulation syndrome (OHSS) by an open labeled, prospective, and randomized clinical trial (RCT) in IHH patients in a single center of the Obstetrics and Gynecology Hospital Affiliated to Fudan University. The onset of patients' mental and psychological diseases such as depression and anxiety rely on their reproductive needs and pregnancy outcomes, which will also be investigated in the current study. Moreover, the effect of clinical interventions to improve pregnancy outcomes and emotional disorders would be discussed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IHH (primary amenorrhea (with or without a history of hormone supplementation therapy); basic LH levels <5IU/L, FSH<5IU/L or normal; no organic lesions in the hypothalamus and pituitary MRI).
* Women of childbearing age who desire to get pregnant

Exclusion Criteria:

* Premature ovarian insufficiency or premature ovarian failure
* Primary amenorrhea due to hypothalamic/pituitary lesions
* Secondary amenorrhea

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women aged between 18-45 years is reproductive. IHH patients in the age have willings to get pregnant and they would seek helps in outpatient clinic of Gynecological endocrinology.
Enrollment: 46 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7 weeks
  Defined as the presence of a gestational sac under ultrasonography
Cumulative pregnancy rate | 12 weeks
  Defined as a pregnancy with a detectable heart rate at 12 weeks of gestation or beyond.
Live birth rate | 42 weeks or beyond
  Defined as the number of deliveries that resulted in a live born neonate, expressed per 100 pregnancies.

SECONDARY OUTCOMES:
Number of IHH patients ending in early pregnancy loss | 12 weeks
  Early pregnancy loss is defined as the loss of a pregnancy prior to 12 weeks gestation
Number of IHH patients with ovarian hyperstimulation syndrome | 12 weeks or beyond
  Ovarian hyperstimulation syndrome is defined as an exaggerated response to excess hormones. It usually occurs in women taking injectable hormone medications to stimulate the development of eggs in the ovaries. Ovarian hyperstimulation syndrome (OHSS) causes the ovaries to swell and become painful.

OTHER OUTCOMES:
Serum progesterone levels on Day 1, 7, and 14 after ovulation | 7 weeks
  Serum progesterone levels is a symbol of luteal function

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Ph.D.,M.D., Principal Investigator — GCP office
Locations (2):
- China (2):
  - OB & GYN Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Obstetrics and Gynecology Hospital of Fudan University, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No